CLINICAL TRIAL: NCT04604652
Title: A Phase 2 Open Label, Proof of Concept Study of HTD1801 (BUDCA) in Adult Subjects With Primary Biliary Cholangitis (PBC) and an Inadequate Response to Standard Therapy - PRONTO-PBC
Brief Title: Open-Label Study of HTD1801 in Adult Subjects With Primary Biliary Cholangitis
Acronym: PRONTO-PBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTD1801.PCT013
Record Dates: First submitted 2020-10-16; First posted 2020-10-27 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-09

CONDITIONS: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; Cholangitis; Cholestasis; Biliary Tract Diseases; Bile Duct Stricture
Keywords: Open-label
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangitis; Cholestasis; Biliary Tract Diseases

STUDY DESIGN:
Intervention Model Description: Single group open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): HTD1801 (BUDCA) 250 mg tablets. Dosed at 1000 mg BID with food.
  Interventions: Drug: HTD1801 (BUDCA)

INTERVENTIONS:
Drug: HTD1801 (BUDCA) — HTD1801 (BUDCA) 250 mg tablets. Dose 1000 mg twice daily with food for 12 weeks.

SUMMARY:
The purpose of this open-label study is to evaluate the safety and tolerability of HDT1801 (BUDCA) over 12 weeks in adult subjects with PBC who have an inadequate response to standard therapy. Inadequate response is defined as persistently elevated serum alkaline phosphatase at greater than or equal to1.5 times the upper limits of normal for the testing lab in spite of having been on adequate doses of standard therapy with UDCA (ursodeoxycholic acid) at 13-15 mg/kg for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of PBC as confirmed by patient history consistent with the American Association for the Study of Liver Diseases (AASLD) Practice Guideline confirmed by two of the following three criteria:

  1. Biochemical evidence of cholestasis with elevation of ALP activity
  2. Presence of antimitochondrial antibody (AMA)
  3. Histopathologic evidence of non-suppurative cholangitis and destruction of small or medium-sized bile ducts if biopsy performed Note: historical AMA and liver biopsy data may be used but must be recorded in source documentation.
* Has been taking a stable, adequate dose of at least (13-15 mg/kg/day) of UDCA for at least 6 months with a serum ALP of at least ≥1.5 × ULN at any time after being on UDCA for >6 months (historical value) and at Screening. If the historical ALP was obtained less than 6 months prior to study start as part of standard of care, the subject may be screened and a second ALP value should be obtained as part of screening, There must be at least a 4-week interval between the ALP values and the ALP values must be ≥1.5 × ULN
* If the subject is taking cholestyramine or other bile acid sequestrant for pruritus, must be on a stable dose no more than once a day for at least 8 weeks prior to Baseline visit. Must be willing and able to take cholestyramine at least 2 hours before or after study medication
* Females of child-bearing potential and males participating in the study must either agree to use at least two approved barrier methods of contraception or be completely abstinent from sexual intercourse, if this is their usual and preferred lifestyle, throughout the duration of the study and for three months after stopping study drug. Females who are postmenopausal must have appropriate documentation
* Able to provide consent

Exclusion Criteria:

* Uncontrolled concomitant autoimmune hepatitis (AIH). Subject should be on no more than 5 mg per day of prednisone (or equivalent dose for other corticosteroids) or no more than 150 mg per day of azathioprine at stable doses and serum ALT should be ≤ 5 × ULN. Enrollment of subjects with controlled AIH will be limited to a total of 5 subjects.
* History of alcohol or substance abuse
* Prior liver transplantation or currently listed for liver transplantation
* History of chronic viral hepatitis, types B or C
* Platelet count ≤150,000/mm3, albumin <3.0 g/dL, International Normalized Ratio (INR) >1.2, or a history of ascites, or encephalopathy, or history of variceal bleeding
* Total bilirubin >1.3 × ULN unless subject has Gilbert Syndrome. If subject has increased total bilirubin due to Gilbert's Syndrome, then direct bilirubin should be <0.3 mg/dL.
* Hemoglobin <10 g/dL for males or females
* Serum TSH level <0.1 or >10 u/mL (subject may be re-screened if hyper- or hypothyroidism has been corrected)
* Renal impairment with eGFR <60 ml/min (CKD stages 3, 4 or 5)
* Human immunodeficiency virus (HIV)-1 or HIV-2 infection by history
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of malignancy within the past 2 years or ongoing malignancy other than basal cell carcinoma, or resected noninvasive cutaneous squamous cell carcinoma
* Active, serious infections that require parenteral antibiotic or antifungal therapy within 30 days prior to Screening
* Major surgical procedure within 30 days of Screening or prior solid organ transplantation
* Females who are pregnant or breastfeeding
* Current or anticipated treatment with radiation therapy, cytotoxic chemotherapeutic agents, and immune-modulating agents (such as interleukins, interferons)
* Diseases that may result in increased serum ALP activities from sources other than the biliary system (e.g., Paget's disease of bone, osteomalacia)
* Allergy to the clinical trial material or its components
* Having received any experimental medications within 28 days prior to Screening
* Use of bezafibrate or fenofibrate within 28 days prior to first day of IP dosing
* Use of obeticholic acid (OCA) within 28 days prior to first day of IP dosing
* Any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing and protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian DiBisceglie, MD, Study Director — HighTide Therapeutics Biopharma Pty.
Locations (12):
- United States (12):
  - University of Miami Schiff Center for Liver Disease, Miami, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health Services, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Northshore University Hospital, Manhasset, New York
  - University GI, Providence, Rhode Island
  - Baylor Research Institute, Dallas, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Liver Institute of Virginia, Newport News, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 46 subjects were screened of which 24 subjects were eligible and enrolled in the study. Subjects discontinued use of ursodeoxycholic acid (UDCA) at baseline prior to transitioning to HTD1801.
Groups:
- HTD1801 1000 mg Twice Daily (BID): All subjects received HTD1801 1000 mg (4 x 250 mg tablets) administered orally twice daily (BID) with food for 12 weeks.
Period: Overall Study
Arm/Group | HTD1801 1000 mg Twice Daily (BID)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HTD1801 1000 mg BID: All subjects received HTD1801 1000 mg (4 x 250 mg tablets) administered orally twice daily with food for 12 weeks.
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Alkaline Phosphatase (ALP) [Mean (Standard Deviation); unit: U/L] | 289.6 (119.8)
Total Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.3)
Gamma-glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: U/L] | 211.0 (187.6)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 216.7 (47.8)
Immunoglobulin M (IgM) [Mean (Standard Deviation); unit: mg/dL] | 340.6 (246.1)
GLOBE score [Mean (Standard Deviation); unit: units on a scale] — The GLOBE score is a validated risk assessment tool providing an estimate of transplant-free survival for patients with PBC. It was developed by the GLOBAL PBC Study Group using Cox regression model on over 4,000 patients with PBC. Lower GLOBE score predicts lower risk. It is calculated using age and levels of ALP, total bilirubin, platelets, and albumin.
  units on a scale | 0.3 (0.7)
Pruritus Visual Analog Scale (VAS; average itch) [Mean (Standard Deviation); unit: cm] — Pruritus VAS is a self-reported instrument for measurement of itch intensity using 24-hour recall period. Subjects were asked to rate the average intensity of their itch on a 10 cm horizontal line ranging from 0 (no itch) to 10 (worst imaginable itch).
  cm | 1.0 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Alkaline Phosphatase (ALP) at Week 12 Compared to Baseline
Description: To evaluate the effects of HTD1801 on serum ALP in adult subjects with PBC who have experienced an inadequate response to standard therapy.
  Inadequate response is defined as ALP ≥1.5 × upper limit of normal (ULN) despite having been on adequate doses of ursodeoxycholic acid (UDCA) for at least 6 months. A reduction in ALP represents an improvement.
Time Frame: Baseline to Week 12
Population: ITT Population: Included all subjects that received at least one dose of HTD1801
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
percent change | -7.7 (23.3)
Statistical Analysis 1: Comparison: HTD1801 1000 mg BID; A t-test was performed to test for the percent change from baseline to Week 12. This analysis was based on observed data without imputation. Testing was one sided using a 5% alpha level. No multiplicity adjustment was used, and the p-values reported for the endpoints were descriptive in nature; Test type: Other; p = 0.077, t-test, 1 sided

2. Secondary Outcome: Change in Total Bilirubin From Baseline to Week 12
Description: To evaluate the effects of HTD1801 on serum markers of cholestasis. A reduction in total bilirubin represents an improvement in a marker of cholestasis.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
mg/dL | -0.10 (0.20)

3. Secondary Outcome: Change in Serum Gamma-glutamyl Transferase (GGT) From Baseline to Week 12
Description: To evaluate the effects of HTD1801 on serum markers of cholestasis. A decrease in GGT represents an improvement in a marker of cholestasis.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
U/L | -34.1 (153.8)

4. Secondary Outcome: Change in Serum Total Cholesterol From Baseline to Week 12
Description: To evaluate the effects of HTD1801 on serum lipids. A reduction in total cholesterol represents an improvement in serum lipids.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
mg/dL | -18.8 (35.1)

5. Secondary Outcome: Change in Immunoglobulin M (IgM) From Baseline to Week 12
Description: To evaluate the effects of HTD1801 on serum markers of inflammation. A reduction in IgM represents an improvement in a marker of inflammation.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
mg/dL | -36.8 (71.4)

6. Secondary Outcome: Change in GLOBE Score Between Baseline and Week 12
Description: The GLOBE score is a validated risk assessment tool providing an estimate of transplant-free survival for patients with PBC. It was developed by the GLOBAL PBC Study Group using Cox regression model on over 4,000 patients with PBC. Lower GLOBE score predicts lower risk. It is calculated using age and levels of ALP, total bilirubin, platelets, and albumin.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
units on a scale | -0.07 (0.3)

7. Secondary Outcome: Change in Pruritus as Measured by Pruritus Visual Analog Score (VAS) From Baseline to Week 12
Description: Pruritus Visual Analog Scale (VAS) is a self-reported instrument for measurement of itch intensity using 24-hour recall period. Subjects were asked to rate the average intensity of their itch on a 10 cm horizontal line ranging from 0 cm (no itch) to 10 cm (worst imaginable itch). A decrease in the Pruritus VAS represents an improvement in itch intensity.
Time Frame: Baseline to Week 12.
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HTD1801 1000 mg BID
Number analyzed (Participants) | 20
units on a scale | -0.9 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 16-week period, including a 12-week treatment period and 4-week followup.
Arm/Group | HTD1801 1000 mg BID
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HTD1801 1000 mg BID (N=24)
COVID-19 Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HTD1801 1000 mg BID (N=24)
Diarrhea (Gastrointestinal disorders) | 9
Abdominal Distension (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2 — 1 subject experienced an adverse event after study drug discontinuation (follow-up period)
Pyrexia (General disorders) | 2 — Adverse events occurred after study drug discontinuation (follow-up period)
Bronchitis (Infections and infestations) | 2 — 1 subject experienced an adverse event after study drug discontinuation (follow-up period)
Upper Respiratory Tract Infection (Infections and infestations) | 2
Liver Function Test Increased (Investigations) | 4 — Adverse events occurred after study drug discontinuation (follow-up period)
Alanine Aminotransferase Increased (Investigations) | 2 — 1 subject experienced an adverse event after study drug discontinuation (follow-up period)
Aspartate Aminotransferase Increased (Investigations) | 2 — 1 subject experienced an adverse event after study drug discontinuation (follow-up period)
Decreased Appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 — 1 subject experienced an adverse event after study drug discontinuation (follow-up period)

LIMITATIONS AND CAVEATS:
This was a small, open-label, proof of concept study with no control group where subjects discontinued UDCA at Baseline. Limitations of the study include potentially being underpowered for the primary endpoint and the safety included adverse events from the 4-week follow-up period after treatment discontinuation. Additional placebo-controlled studies are needed to further evaluate the benefit of HTD1801 in PBC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT04604652/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04604652/SAP_001.pdf